CLINICAL TRIAL: NCT05432687
Title: Impact de l'incompétence Abdominale Sur l'Icontinence Urinaire Post Prostatectomie
Brief Title: Impact of Abdominal Incompetence on Urinary Incontinence After Prostatectomy (PROSTABDO)
Acronym: PROSTABDO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021/664
Record Dates: First submitted 2022-06-13; First posted 2022-06-27 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient before Robotic-assisted Radical Prostatectomy (Other): evaluation of deep abdominal wall before surgery : cough test + ulstrasonography of transversus abdominis
  Interventions: Diagnostic Test: evaluation of deep abdominal wall before surgery

INTERVENTIONS:
Diagnostic Test: evaluation of deep abdominal wall before surgery — : cough test (L guillarme) + ulstrasonography of transversus abdominis

SUMMARY:
the aim of this study is assess deep abdominal wall (ultrasonography of transversus abdominis muscle) before prostatectomy, and look at one year post surgery if patient with several incontinence are the same who have dysfunction (abdominal incompetence) before the surgery.

ELIGIBILITY:
Inclusion Criteria:

* male with prostate cancer going to have a robotic-assisted laparoscopic radical prostatectomy

Exclusion Criteria:

* neurological patology with bladder impact (SCI, parkinson disease, multiple sclerosis....)
* urinary incontinence before surgery
* surgery for abdominal wallhernia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
amount of incontinence after surgery (1 year) | 1 year
  mesured with pad test on 3 days

SECONDARY OUTCOMES:
amount of incontinence after 3 month | 3 month
  mesured with pad test on 3 days
amount of incontinence after 6 month | 6 month
  mesured with pad test on 3 days
quality of life after 3 month | 3 month
  Short-Form (SF-36) Health Survey
quality of life after6 month | 6 month
  Short-Form (SF-36) Health Survey
quality of life after 12 month | 12 month
  Short-Form (SF-36) Health Survey
quality of incontinence after 12 month | 12 month
  mesured with urinary symptom profil score

CONTACTS AND LOCATIONS:
Overall Officials: Emilie CERUTTI, Principal Investigator — University hospital of Besançon
Locations (1):
- University hospital of Besançon, Besançon, France